CLINICAL TRIAL: NCT06867900
Title: Unexplained Recurrent Pregnancy Loss: New Therapeutic Perspectives
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1355
Record Dates: First submitted 2023-07-06; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-09

CONDITIONS: Miscarriage, Recurrent
Keywords: Recurrent pregnancy loss
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bifidobacterium Longum (Experimental)
  Interventions: Dietary Supplement: Bifidobacterium Longum ES1

INTERVENTIONS:
Dietary Supplement: Bifidobacterium Longum ES1 — Oral administration of Bifidobacterium Longum ES1 for three months.

SUMMARY:
Evaluation of gut permeability and endometrial inflammasome NLRP3 in women with unexplaid recurrent pregnancy loss before-after administration of Bifidobacteriumlongum ES1.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic recurrent pregnancy loss
* Genetic predisposition to celiac disease

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2025-07-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of Endometrial inflammation in RPL women | 3 months
  Analysis of the inflammasome NALP3 expression and activation in serum and endometrial fluid in women with unexplained recurrent pregnancy loss compared to women with uncomplicated pregnancy history.
Assessment of Gut permeability status in RPL women | 3 months
  Analysis of zonulin expression and activation in serum and endometrial fluid in women with unexplained recurrent pregnancy loss compared to women with uncomplicated pregnancy history.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Tersigni, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Reasearch Laboratory 3J IRCCS Gemelli, Rome, Italy